CLINICAL TRIAL: NCT07178990
Title: Mobile Platform for Optimizing Wellness and Engagement in Recovery
Acronym: MPOWER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); DynamiCare Health (Industry)
Responsible Party: Principal Investigator, Anne Fernandez, Associate Professor of Psychiatry, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00266546; 1R34AA031870-01 (NIH)
Record Dates: First submitted 2025-09-10; First posted 2025-09-17 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Opioid Agonist Treatment; Alcohol Use Disorder; Opioid Use Disorder
Keywords: Research surveys; App based program; Smartphone
MeSH Terms: conditions — Alcoholism; Opioid-Related Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Contingency Management (CM) Intervention Arm (Experimental): After participants meet eligibility and complete the DynamiCare assessment period, participants randomized to this group will receive a comprehensive digital CM platform designed to enhance OAT retention and promote abstinence from alcohol and opioids. This will include the DynamiCare Motivation Support Program.
  Interventions: Behavioral: Digital Contingency Management Intervention Arm
- Wellness Condition (Active Comparator): After participants meet eligibility and complete the DynamiCare assessment period, those randomized to this group will receive a wellness digital platform that includes surveys, testing, and tech support.
  Interventions: Behavioral: Digital Wellness Arm

INTERVENTIONS:
Behavioral: Digital Contingency Management Intervention Arm — Participants will use a version of the app for 6-months. Participants in this group may earn rewards for completing recovery-related activities and for abstinence from drugs and alcohol. During the 6 months this will include: random saliva drug tests, breathalyzer tests, and video selfies, completing surveys and questionnaires through the app, and receiving rewards on a debit card for abstinent tests, surveys, and activities. Additionally, participants will complete follow-up at approximately 9 months after randomization.
  Arms: Digital Contingency Management (CM) Intervention Arm
Behavioral: Digital Wellness Arm — Participants will use a version of the app for 6-months focussed on wellness. During the 6 months this will include: random requests to do saliva drug tests, breathalyzer tests, and video selfies, complete surveys and questionnaires through the app, and receive rewards on a debit card for completing tests, surveys, and activities. Participants in this group may also earn rewards for completing study activities like tests and surveys. Additionally, participants will complete follow-up at approximately 9 months after randomization.
  Arms: Wellness Condition

SUMMARY:
This pilot study addresses the urgent public health crisis of co-occurring opioid and alcohol use disorders (OUD-AUD), leading causes of mortality in the United States, by testing a scalable digital contingency management (CM) treatment among Medicaid beneficiaries. The study aims to evaluate the feasibility and acceptability of digital CM for OUD-AUD recovery, while also planning for broader implementation.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be enrolled in the Michigan Medicaid program
* Opioid agonist treatment (OAT): Participants must have initiated OAT with buprenorphine or methadone
* Participants must have an OAT prescription and Alcohol use disorder (AUD) based on self-report measure during screening
* Participants must have regular access to a working smartphone and internet connection.
* Participants must have a reliable mailing address to receive study supplies (e.g., salivary drug tests).

Exclusion Criteria:

* Primary Medicare Coverage: Individuals that are dual-eligible for Medicaid and Medicare and aged 65 or older, due to limited availability of Medicaid claims data for this group
* Individuals that cannot voluntarily provide informed consent themselves for any reason, including legal incompetency
* Individuals with substantial cognitive impairment that would interfere with study participation
* Individuals unable to read or understand English
* Individuals experiencing active suicidality or psychosis.
* Individuals with a planned admission to residential treatment or incarceration during the study period.

Ages: 19 Years to 63 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility based on recruitment | Recruitment period 12 months
  Recruitment: ≥60% of participants enrolled
Feasibility based on adherence | 6 months (during the Dynamicare program)
  Adherence: ≥50% of app-based, biochemically-verified tests completed in the digital CM condition.
Feasibility based on Retention | 6 months
  Retention: ≥70% of participants retained at 6 months
Acceptability of the intervention | 3-month after starting program
  Defined as >70% of participants rating the intervention experience ≥ 4/5 on the Acceptability of Intervention Measure

CONTACTS AND LOCATIONS:
Overall Officials: Anne Fernandez, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
National Institute on Alcohol Abuse and Alcoholism (NIAAA)-funded investigators conducting applicable human subjects research are expected to submit de-identified, individual-level data to this data archive. The data generated in this grant will also be presented at national or international meetings (e.g., Research Society on Alcoholism, Addiction Health Services Research, etc.) and published in a timely fashion. All final peer-reviewed manuscripts that arise from this proposal will be submitted to the digital archive in PubMed Central.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The research team will share data with NIAAA data archive (NIAAADA) biannually per funder requirements. The data in the NIAAADA are catalogued and made available to the general research community at the time of an associated publication or end of the award/support period, whichever comes first. Data in the NIAAADA is available indefinitely.
Access Criteria: Community of scientists interested in the study of alcohol use and related interventions. Additionally, data submitted to National Institute on Alcohol Abuse and Alcoholism Data Archive (NIAAADA) will be accessible by the general research community via NIAAADA.
URL: https://nda.nih.gov/niaaa